CLINICAL TRIAL: NCT01030562
Title: Immunogenicity of the HPV-6, 11, 16, 18 Vaccine Among Adolescent Girls Who Receive Vaccine Doses at Non-recommended Intervals and Factors Related to Non-adherence
Brief Title: Immunogenicity of Off-Schedule Dosing of HPV Vaccine
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 08-0012
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2013-07-31

CONDITIONS: Papilloma Viral Infection
Keywords: adolescent; children; HPV; human papillomavirus; vaccine; women
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Serum samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Alternate Arm: Subjects who meet eligibility requirements but do not fit into any of the primary experimental arms.
- Control Arm: Subjects with an on-time interval between Dose 1 and 2 and an on-time interval between Dose 2 and 3.
- Experimental/Primary Arm 1: This primary arm will consist of subjects receiving the second dose on time/third dose substantially late.
- Experimental/Primary Arm 2: This primary arm will consist of subjects receiving the second dose substantially late/third dose on time.
- Experimental/Primary Arm 3: This primary arm will consist of subjects receiving the second dose substantially late/third dose substantially late.

SUMMARY:
The purpose of this study is to gain a better understanding of the body's response to a human papillomavirus (HPV) (sexually transmitted disease), vaccine and booster shot. The study will also determine factors related to adolescents not following vaccination schedules. The HPV vaccine requires 3 doses (shots). Girls sometimes receive the 3 shots at the recommended time and sometimes girls receive the shots at non-recommended times. This study will evaluate if getting the shots at non-recommended times affects the level of protection provided by the vaccine. Participants will include about 1400 girls 9-17 years old receiving a third dose of HPV vaccine from their primary care clinician. The parent/legal guardian of each subject may answer a questionnaire related to the vaccine schedule. Study procedures include: medical history, questionnaires and blood draws. Participants will be involved in the study for about 6 months from time of enrollment.

DETAILED DESCRIPTION:
The immune response to the quadrivalent human papillomavirus (HPV) vaccine in the non-clinical trial settings is unknown. In addition, the immune response following administration of vaccine at substantially prolonged intervals is unknown. Early indications suggest that many girls will be receiving the vaccine at prolonged intervals and that this timing may affect immunogenicity. The lack of knowledge about the immunogenicity of prolonged intervals between vaccine doses precludes evidence based recommendations for patients who are substantially late for their second or third dose. Some clinicians currently restart the series while others give the doses at the incorrect interval (unpublished observation) without the ability to counsel their patients as to their expected level of immune response or protection. Examining the immune response prior to the third dose and at one and six months after the third dose will allow a better understanding of the immunogenicity of this vaccine and immune response to booster doses. Furthermore, determining factors related to non-adherence in the adolescent age group is important and timely. As an increasing number of vaccines are being recommended to the adolescent age group, elucidating factors involved with non-adherence to the recommended dosing schedule is now critical. This information can guide interventions that aim to increase adolescent adherence to the recommended schedules. Eligible girls 9 - 17 years old receiving the quadrivalent HPV vaccine from their primary care provider will be enrolled into this study on the day of, but prior to, receiving their third HPV vaccine dose or at approximately 28 days after the third HPV dose . Blood for immunogenicity testing will be obtained up to three times throughout the study: one month (Study Day 28) and six months (Study Day 180) after the third dose (Study Day 0) for all subjects and just prior to the third dose for subjects on time for their third dose (regardless of the time interval between the first and second dose). The primary analysis will be based on comparing the geometric mean titer (GMTs) and sero-response rate of subjects receiving the vaccine doses at substantially prolonged intervals to GMTs and sero-response rate of subjects receiving the second and third dose on time. In addition, on Study Day 0, patient and parent related factors known to impact health care utilization may be measured using a questionnaire given to parents/legal guardians and 14 to 17 year old subjects. Analysis based on a health care utilization model will be used to determine factors associated with non-adherence to the vaccine schedule. Initially, all subjects meeting eligibility criteria will be enrolled regardless of timing of the second and third vaccine doses. When a study arm reaches the accrual target, it will be closed to enrollment. Enrollment for the entire study will remain open until the control and three primary experimental arms have completed enrollment One or more experimental arms may be dropped from the study after monitoring of accrual rates indicates that it/they cannot be fully enrolled in a timely fashion. Monitoring will occur monthly. Assessment of accrual rates will occur semi-annually. The primary objective is to compare the GMT one month after completing the three dose vaccination series in 9 to 17 year old subjects who received the second and/or third dose at substantially prolonged intervals to subjects who receive both the second and third dose on time after adjusting for age.

ELIGIBILITY:
Inclusion Criteria:

Girls will be eligible if they are: -9 to 17 years of age (defined as between 9 years 0 days and younger than 18 years of age) at time of receipt of third HPV dose; -Receiving the third human papillomavirus (HPV) vaccine as part of routine health care; -Able and willing to complete all study visits and evaluations; -Able and willing to participate in the study by providing written informed assent/consent (as applicable); -Parent or legal guardian provides permission (as applicable). Parent/legal guardian inclusion criteria: At sites administering the survey and health literacy assessment, parent or legal guardian providing permission for their daughter to participate in the study will be eligible to participate in the parental questionnaire if they are able to provide informed consent for themselves.

Exclusion Criteria:

Girls meeting any of the following exclusion criteria at baseline will be excluded from study participation. -Unable to comply with the study protocol. -Receipt of more than 3 doses of human papillomavirus (HPV) vaccine. -Receipt of blood and or blood products (including immunoglobulin) in the past 3 months or anticipated receipt during the study period. -History of any physical, mental, or developmental disorder that study personnel believe may hinder a participant's ability to comply with the study requirements. -History of malignancy or confirmed or suspected immunodeficient condition, such as human immunodeficiency virus infection. -Receipt of or history of receipt of any medications or treatments that affect the immune system, such as immune globulin, interferon, immunomodulators, cytotoxic drugs or other drugs known to be frequently associated with significant major organ toxicity since six months prior to the first HPV vaccine dose. -Receipt of long-term (greater than or equal to 2 weeks) potentially immunosuppressive corticosteroid use within six months or anticipated receipt during the study period. Specifically, potentially immunosuppressive corticosteroids or any parenteral corticosteroid, high dose (>800 mcg/day) beclomethasone dipropionate or equivalent medication; nasal and topical steroids are allowed. -Current or former participation in HPV vaccine related research. -Receipt of an investigational or alternate (Cervarix) HPV vaccine. -Receipt of a live virus vaccine (varicella virus vaccine, any measles, mumps, or rubella virus vaccine, or yellow fever vaccine but not including live attenuated influenza virus vaccine) within 4 weeks before or after the 3rd dose of HPV vaccine or anticipated receipt of a live virus vaccine within 4 weeks after the 3rd dose of HPV vaccine. However, subjects may receive any vaccine on the same day as the third dose of HPV. Parent/legal guardian exclusion criteria: If the site is actively recruiting adolescents from a clinic population, the survey and health literacy assessments are not available for the parents/legal guardians from that clinic population. Therefore they will not be asked to participate in the study. -At sites administering the survey and health literacy assessment, parents/legal guardians meeting any of the following exclusion criteria at baseline will be excluded from filling out the study questionnaire examining factors associated with adherence: -History of any physical, mental or developmental disorder that study personnel believe may hinder a participant's ability to comply with study requirements.

Ages: 9 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Girls 9-17 years old receiving third dose of HPV vaccine from primary care clinician. Parent/legal guardian will participate by answering a questionnaire to determine factors related to non-adherence to recommended vaccine schedule.
Sampling Method: Non-Probability Sample
Enrollment: 1321 (Actual)
Dates: Start 2010-06-02 (Actual); Primary Completion 2014-03-05 (Actual); Study Completion 2014-03-05 (Actual)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) to vaccine human papillomavirus (HPV) serotypes as measured by HPV4-plex IgG ELISA. | One month after the third HPV vaccine dose.
Sero-response rate (proportion of subjects developing antibody to vaccine HPV serotypes). | One month after the third HPV vaccine dose.

SECONDARY OUTCOMES:
GMT to vaccine HPV serotypes as measured by HPV4-plex IgG ELISA | Prior to the third HPV vaccine dose and six months after the third HPV vaccine dose.
Sero-response rate (proportion of subjects developing antibody to vaccine HPV serotypes). | Prior to the third HPV vaccine dose and six months after the third HPV vaccine dose.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Kaiser Permanente Crescent Medical Center - Pediatrics/Adolescent Medicine, Tucker, Georgia
  - University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland
  - Children's Mercy Hospital and Clinics - Infectious Diseases, Kansas City, Missouri
  - Cincinnati Children?s Hospital Medical Center - Adolescent Medicine, Cincinnati, Ohio
  - Primary Physicians Research Inc. - Pittsburgh, Pittsburgh, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt - Adolescent Medicine, Nashville, Tennessee
  - Kaiser Permanente Washington Health Research Institute - Vaccines and Infectious Diseases, Seattle, Washington

REFERENCES:
- [Derived] Widdice LE, Hoagland R, Callahan ST, Kahn JA, Harrison CJ, Pahud BA, Frey SE, Berry AA, Kotloff KL, Edwards KM, Mulligan MJ, Sudman J, Nakamura A, Bernstein DI. Caregiver and adolescent factors associated with delayed completion of the three-dose human papillomavirus vaccination series. Vaccine. 2018 Mar 7;36(11):1491-1499. doi: 10.1016/j.vaccine.2017.12.060. Epub 2018 Feb 7. PMID 29428177